CLINICAL TRIAL: NCT06348446
Title: Tacrolimus Exposure and Outcomes in Kidney Transplant Patients: A Retrospective Multicenter Study of Clinical Data Warehouse (CDW) in South Korea
Brief Title: Tacrolimus Exposure in Kidney Transplantation
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: FY20-2963
Record Dates: First submitted 2024-03-24; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Kidney Transplant Rejection
Keywords: kidney transplantation; tacrolimus; acute rejection; graft survival; adverse event

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Using CDW data from 5 tertiary hospitals in Korea, this study identify the optimal range of trough level that can prevent adverse outcome in the early periods after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients between January 1, 2005 through December 31, 2014 in one of the five participating centers
* Patients receiving oral tacrolimus as one of the main immunosuppressant at the start of the defined cohort time (i.e. at post-transplant 2 months for the analysis of 1-year outcomes and at post-transplant 12 months for the analysis of 6-year outcomes)

Exclusion Criteria:

* Graft failure occurring within the first 2 month of transplantation
* Mortality of any cause occurring within the first 2 month of transplantation
* Patients moving centers during the study period
* Patients who have received other organ transplantation(s) besides renal transplantation in the defined period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All renal transplant recipients between January 1, 2005 through December 31, 2014 in one of the five participating centers are included. Further selection will be undertaken to include only patients receiving oral tacrolimus as one of the main immunosuppressant at post-transplant 2 month (for early outcomes) and post-transplant 1 year (for late outcomes).
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
relationship between time varying periodic mean of tacrolimus trough and a composite 1-year allograft outcomes | 1 year after transplantation
  the relationship between time varying periodic mean of tacrolimus trough level during 2-12 mo. post-transplant and a composite of 1-year allograft outcomes consisting of biopsy proven acute rejection, renal dysfunction (eGFR<30), development of dnDSA, and death censored graft failure that occurred within 1 year from the latest transplant.

SECONDARY OUTCOMES:
relationship between time varying periodic mean of tacrolimus trough level during 12-72 mo. post-transplant and 6-year composite allograft outcome | 6 year after transplantation
  the relationship between time varying periodic mean of tacrolimus trough level during 12-72 mo. post-transplant and 6-year composite allograft outcome that occurred within 6 years from the latest transplant
relationship between post-transplant time varying periodic mean tacrolimus trough level and severe infection | 6 year after transplantation
  the relationship between post-transplant time varying periodic mean tacrolimus trough level and severe infection (1-year and 6-year)
relationship between post-transplant time varying periodic mean tacrolimus trough level and cardiovascular event | 6 year after transplantation
  the relationship between post-transplant time varying periodic mean tacrolimus trough level and cardiovascular event (1-year and 6-year)
relationship between post-transplant time varying periodic mean tacrolimus trough level and patient mortality | 6 year after transplantation
  the relationship between post-transplant time varying periodic mean tacrolimus trough level and patient mortality (1-year and 6-year)

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Asan medical center, Seoul, Korea, Seoul
  - Samsung medical center, Seoul, Korea, Seoul
  - Seoul St. Mary's hospital, Seoul, Korea, Seoul
  - Severance hospital, Seoul, Korea, Seoul

IPD SHARING:
Plan to Share IPD: Undecided